CLINICAL TRIAL: NCT03300986
Title: Parameter Changes in Functional Electrical Stimulation
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: MP16/017
Record Dates: First submitted 2017-08-11; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Gait Disorders, Neurologic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Functional Electrical Stimulation (FES) users

SUMMARY:
This study aims to look at how changes to a person's functional electrical stimulation might change how they walk. Functional electrical stimulation (FES) is commonly used to help people with foot drop from upper motor neurone conditions such as stroke or multiple sclerosis. This group of people have muscle weakness which makes it difficult to lift the foot, which causes trips and falls.

FES reduces foot drop by using a portable device to apply short electrical pulses to the nerve which lifts the foot. The FES device stimulates this nerve only during the swing phase, when the foot is off the floor. Typically this is achieved by using a foot-switch, which detects when the heel leaves the floor. Stimulation begins a short interval of time after the heel leaves the floor, ramps up from zero to set stimulation for the individual, and at another period of time after the heel hits the floor, stimulation ramps down from set amount to zero. There are four time intervals described here which can be varied by the clinician on the device:-

* Delay (the time between heel lift and the start of stimulation)
* Ramp up (the time for stimulation to reach full strength)
* Extension (the time between heel strike and the ramp down)
* Ramp down (the time for stimulation to reach zero from full strength) These intervals are usually set by experienced clinicians using a qualitative assessment of the patient's walking and trial-and-error. A literature review has found no published studies which compare walking with different timing. This knowledge would be useful for clinicians, who could use this information as a starting point in finding the best timing parameters for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Upper motor neurone lesion causing foot drop
* Currently use single-channel Odstock Medical ODFS functional electrical stimulator
* Age 18 or older
* Attending Leeds FES Service follow-up clinics

Exclusion Criteria:

* • FES user for less than three months

  * Lower limb prosthesis
  * Cannot walk 5m with walking aids
  * Cannot walk twenty 5m walks within a three-hour period
  * Use FES less than once per week

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population for this study is adult users of standard FES for foot drop, registered with the Leeds FES service. Any upper motor neurone lesion can be the primary condition.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Gait analysis will be measured according to routine protocol | Gait will be assessed over one visit of three hours.
  Gait analysis will measured in accordance with the Plug-In-Gait model guide. This measures 16 points on the subjects left and right leg.